IRAS Project ID: 351521

**Version**: 1 (02-04-25)

Title: The Effect of PMPR and Chlorhexidine Mouthwash on Salivary and Acquired Enamel Pellicle (AEP) Proteins and Vascular Function and Inflammation in People with Periodontal Disease.

Chief Investigator: Saagarika Sharma
William Beatty Building,
Faculty of Science and Health,
School of Dental, Health and Care Professions,
University of Portsmouth
PORTSMOUTH,
PO1 2QG

Telephone: 02392 84 5528

Email: <a href="mailto:saagarika.sharma@port.ac.uk">saagarika.sharma@port.ac.uk</a>



William Beatty Building, School of Dental, Health and Care Professions, University of Portsmouth, PORTSMOUTH, PO1 2QG, UK

## **CONSENT FORM**

NHS REC Reference No: 25/WA/0160

Title of Project: The Effect of PMPR and Chlorhexidine Mouthwash on Salivary and Acquired Enamel Pellicle (AEP) Proteins and Vascular Function and Inflammation in People with Periodontal Disease

Name and Contact Details of Researcher(s): Saagarika Sharma

Email:saagarika.sharma@port.ac.uk

+44(0) 23 9284 5528

Name and Contact Details of Supervisor (if relevant):

Data Protection Officer: Samantha Hill, 023 9284 3642 or information-matters@port.ac.uk Ethics Committee Reference Number:

- I confirm that I have read and understood the information sheet dated 02-04-25 (version 1) for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily.
- 2. I understand that my participation in this research study is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected.

## IRAS Project ID: 351521

**Version**: 1 (02-04-25)
Title: The Effect of PMPR and Chlorhexidine Mouthwash on Salivary and Acquired Enamel Pellicle (AEP) Proteins and Vascular Function and Inflammation in People with Periodontal Disease.

| 3. | I understand that data collected during this study will be processed in accordance with data protection | |
|---|---|---|
| | law as explained in the Participant Information Sheet. | |
| 4. | I understand that the data/saliva/blood samples collected up to the point of withdrawal or losing | |
| | capacity will be retained. | |
| 5. | I understand that I am also providing consent for the collection of samples and measurements | |
| | related to vascular health, including blood pressure monitoring, ultrasound assessments, and | |
| | evaluations of artery function. | |
| 6. | I understand that the results of this study may be published and/or presented at meetings or academic | |
| | conferences and may be provided to research commissioners. I give my permission for my anonymous | |
| | data, which does not identify me, to be disseminated in this way. The collected data from this study will | |
| | be published in accordance with principles of open access to ensure transparency and widespread | |
| | availability of our findings | |
| 7 | I agree that the data from this study will be shared with sponsor representatives who may see data in an | |
| | identifiable form for monitoring purposes. | |
| | dentification for mornitoring purposess. | |
| 0 | I agree to take part in the above study | |
| ο. | agree to take part in the above study | |
| Optional: Please select one option by marking either "Yes" or "No" in response to the following statement: | | |
| 9. | I agree to the data I contribute to this study being retained for any future research Yes | NO |
| | that has been given a favourable opinion by a Research Ethics Committee, and that | |
| | any retained data will be stored in an anonymised format. | |
| Name of Participant: Date: Signature: | | |
| Na | nme of Researcher: Date: Signature: | |

**Note**: When completed, one copy to be given to the participant, one copy to be retained in the study file by the researcher.